CLINICAL TRIAL: NCT00584337
Title: Coronary CT Angiography as the Primary Initial Method of Evaluating Patients With Subacute Chest Pain (CT PRIME)
Acronym: CTPRIME
Status: Withdrawn | Type: Observational
Why Stopped: It was decided to not proceed with the study at this time.
Sponsor: Corewell Health East (Other)
Responsible Party: Aiden Abidov MD, PhD, Division of Cardiology, William Beaumont Hospital
Other Study IDs: 2007-091
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Artery Disease
Keywords: tomography; coronary artery disease; Stress Test; Coronary CT Angiography; Diagnostic Accuracy; Non invasive testing
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
This study is designed to evaluate a new approach to the diagnosis of chronic or sub-acute chest pain patients in the out-patient setting. Patients in this study are selected to be "low-risk", meaning they are not having an acute or recent heart attack (AMI), based on screening blood tests and electrocardiograms (EKGs). In addition, these patients have a low or intermediate pre-test likelihood of the coronary artery disease (CAD), which means that probability of the CAD based on the available clinical and historical information, does not make a diagnosis of the CAD a certain clinical diagnosis in the particular patient and this, in turn, requires an additional diagnostic work up.

DETAILED DESCRIPTION:
To compare and contrast the diagnostic efficacy of coronary CT angiography (CCTA) to standard of care-myocardial perfusion imaging (MPI) as an initial diagnostic test for evaluation of patients with suspected angina pectoris and no known CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Non-acute (onset≥72 hours) chest pain suggestive of possible underlying CAD in out-patient.
2. Low or low-to-intermediate clinical likelihood of the CAD.
3. Very low or low risk Goldman-Reilly risk group.
4. Ability to provide informed consent.
5. Age equal to or greater than 18 years.

Exclusion Criteria:

1. Intermediate or higher risk of ACS by Goldman-Reilly criteria:

   1. Electrographic evidence of acute ST elevation myocardial infarction (STEMI) with ST segment elevation equal to or greater than 1mm in two or more contiguous leads).
   2. Electrocardiographic evidence of acute non-ST infarction (NSTEMI) or acute myocardial ischemia, including flat to down sloping ST segment depression equal to or greater than 1mm and/or T wave inversion equal to or greater than 2mm in 2 or more leads.
   3. Positive cardiac biomarkers (troponin and/or creatinine phosphokinase MB fraction) compatible with acute myocardial infarction on initial laboratory testing, based on the local laboratory upper range of normal.
   4. Clinical instability including cardiogenic shock, hypotension (systolic blood pressure < 90 mmHg), refractory hypertension (systolic blood pressure > 180 mmHg on therapy), sustained ventricular or atrial arrhythmia requiring intravenous medications.
2. Presence of known pre-existing coronary artery disease (known prior myocardial infarction, EKG evidence compatible with prior infarction, prior angiographic evidence of significant coronary artery disease, history of prior coronary revascularization).
3. Presence of signs or symptoms compatible with obvious non-cardiac chest pain, including musculoskeletal, gastrointestinal or neuropathic causes.
4. Renal insufficiency (creatinine >1.5) or history of chronic or transient renal failure.
5. Atrial fibrillation or other markedly irregular rhythm.
6. Pregnancy or unknown pregnancy status.
7. Known allergy to iodinated contrast.
8. Inability to tolerate beta-blocking drugs, including patients with reactive airways disease requiring maintenance inhaled bronchodilators or steroids, complete heart block or second-degree atrioventricular block.
9. Iodinated contrast administration within the past 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers over 18 years of age; both genders; referred from participating cardiologist's offices
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Primary outcome variable: diagnostic efficiency. | 6 months, 1 year

SECONDARY OUTCOMES:
Secondary outcome variables: diagnostic accuracy, prognostic accuracy. | 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aiden Abidov, MD, PhD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States